CLINICAL TRIAL: NCT06183775
Title: Functional Magnetic Resonance Imaging Study on the Role of Awareness in Visual Perception in Healthy Adult Subjects.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: VISCON-01
Record Dates: First submitted 2023-12-12; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Magnetic Resonance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study concerns the investigation of the role of awareness in visual perception, highlighting the brain systems involved during non-processing Aware of stimuli belonging to different semantic categories. Specifically, the theoretical perspective of reference is that of the so-called "grounded cognition", according to which the representation of the concepts of semantic knowledge is conveyed by information sensorimotor and affective, introspective and social states. The main objective is therefore to evaluate whether the meaning of the stimulus can be extracted in the absence of awareness, investigating the neural response in the brain regions known to be involved in the conscious processing of stimuli belonging to the semantic categories in question.

To this end, two different experimental paradigms were implemented. A first paradigm aimed at investigating the unconscious representation of semantic knowledge in the context of language, therefore using visual stimuli in lexical mode (words). A second paradigm aimed at investigating the same phenomena in the field of visual perception of objects in space, using stimuli in iconic mode (images).

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 65;
* Italian mother tongue.

Exclusion Criteria:

* clinical evidence of significant psychiatric or systemic neurological pathologies.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers, enlisted among the students and workers of the San Raffaele Hospital and other universities.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging for 62 healthy volunteers for measure the role of consciousness in visual perception. | 2 years
  The role of consciousness in visual perception, highlighting the brain areas involved during the processing of stimuli belonging to different semantic categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No